CLINICAL TRIAL: NCT01968096
Title: The Reversal of Neuromuscular Adaptation in Human With Spinal Cord Injury II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Ya-Ju Chang, Associate Professor, Chang Gung University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 102-1780C; NSC102-2314-B-182-021-MY2
Record Dates: First submitted 2013-10-16; First posted 2013-10-23 (Estimated); Last update posted 2013-10-23 (Estimated); Status verified 2013-10

CONDITIONS: Spinal Cord Injury(SCI)
Keywords: Reflex; Post activation; Spinal cord injury; Pre-synaptic inhibition; Machine driven passive strech
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- SCI subjects (No Intervention): Stage 1 subjects: pilot study:understand post activation depression with spinal cord injury to avoid the influence of the suprasegmental level.
- Incomplete SCI subjects (No Intervention): Stage 2 subjects: pilot study:The strength of depression will be evaluated in individuals with and without SCI.
- Health subjects (No Intervention): Stage 2 subjects: pilot study:The strength of depression will be evaluated in individuals with and without SCI.
- SCI subjects with high muscle tone (High frequency) (Experimental): Stage 3 subjects:A rehabilitation program of machine driven passive stretch(High frequency) will be executed .
  Interventions: Device: home-based ankle continuous passive motion machine.
- SCI subjects with high muscle tone(low frequency) (Experimental): Stage 3 subjects:A rehabilitation program of machine driven passive stretch(Low frequency) will be executed.
  Interventions: Device: home-based ankle continuous passive motion machine.
- SCI subjects with high muscle tone (No Intervention): Stage 3 subjects:Control subjects

INTERVENTIONS:
Device: home-based ankle continuous passive motion machine. — A rehabilitation program of machine driven passive stretch.
  Arms: SCI subjects with high muscle tone (High frequency); SCI subjects with high muscle tone(low frequency)

SUMMARY:
Following injury to the spinal cord, the spinal circuit undergoes a series of adaptations. In parallel with the spinal circuit adaptation, the muscular properties also adapt. In human and animal studies, histochemical and physiological evidences showed that the paralyzed muscle transferred from slow, fatigue-resistant to fast, fatigable after injury.

Reversal of neuromuscular property for persons with SCI needs to be resolved. Studies using high load electrical stimulations showed a reverse change of muscular properties, such as hypertrophy and reversal of fiber type transformations but failed to show a reversal of spinal circuitry function. Previous studies found that fast continuous passive motion (CPM) altered the H reflex excitability in human. Animal studies found that passive cycling and passive stretching delayed atrophy and influenced the transition of type I and IIa MHC. Theses findings lead to a hypothesis that mechanical stimulation might be able to reverse both spinal circuitry and muscular properties after SCI but it has not been confirmed in human study.

The purpose of this project is to investigate the effect of mechanical stimulation by fast CPM on the reversing adaptation of human paralyzed muscle after SCI.

ELIGIBILITY:
Stage 1 subjects: Spinal cord injury subject

Inclusion Criteria:

* Clinical diagnosis of spinal cord injury < 2 years

Stage 2 subjects: Incomplete spinal cord injury subject

Inclusion Criteria:

* Clinical diagnosis of incomplete spinal cord injury
* ASIA classification:B, C, or D

Stage 3 subjects: Spinal cord injury subjects with high muscle tone

Inclusion Criteria:

* Clinical diagnosis of spinal cord injury.
* ASIA classification: A, B, C, or D

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Clinical muscle tone tests & Peripheral nerve Stimulation machine | Participants will be followed for the duration of invention, an expected average of 24 weeks.
  Clinical muscle tone test include Modified Ashworth Scale, Pendulum test ,and withdraw reflex,etc.. Normalization of muscle tone, and influence of muscle property will be evaluated.
  Peripheral nerve Stimulation machine stimulate Soleus and Tibialis anterior. Restoration of post activation will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan